CLINICAL TRIAL: NCT06470178
Title: A Real-World Study of Neoadjuvant/Conversion Therapy for Locally Advanced or Metastatic Colorectal Cancer With Chemotherapy Combined With Anti-Angiogenic Targeted Agents
Brief Title: A Real-World Study of Neoadjuvant/Conversion Therapy for Colorectal Cancer With Chemotherapy And Anti-Angiogenic Targeted Agents
Status: Not yet recruiting | Type: Observational
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Bin Xiong, MD, Chief Physician, Wuhan University
Other Study IDs: HMPL-013-C2-CRC09
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer
Keywords: Fruquintinib; anti-angiogenic targeted therapies; colorectal cancer; neoadjuvant therapy; conversion therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 : neoadjuvant treatment
  Interventions: Combination Product: corhot1: chemotherapy combined with fruquintinib
- Cohort 2:conversion treatment
  Interventions: Combination Product: corhot2: chemotherapy combined with fruquintinib

INTERVENTIONS:
Combination Product: corhot1: chemotherapy combined with fruquintinib — Chemotherapy Drugs: Selection based on clinical guidelines/indications and patient condition.For example, recommended chemotherapy regimens: mFOLFOX6 or CAPEOX.
  Fruquintinib: 3mg (starting dose), PO (once daily). Dosing schedule and dosage can be adjusted based on concurrent chemotherapy and immune checkpoint inhibitors. Have received fruquintinib treatment for at least 2 cycles.
  Groups: Cohort 1 : neoadjuvant treatment
Combination Product: corhot2: chemotherapy combined with fruquintinib — Chemotherapy Drugs: Selection based on clinical guidelines/indications and patient condition.For example, recommended chemotherapy regimens: mFOLFOX6 or CAPEOX.
  Fruquintinib: 3mg (starting dose), PO (once daily). Dosing schedule and dosage can be adjusted based on concurrent chemotherapy and immune checkpoint inhibitors. Have received fruquintinib treatment for at least 2 cycles.
  Groups: Cohort 2:conversion treatment

SUMMARY:
Fruquintinib is already the standard third-line treatment for metastatic colorectal cancer, but the efficacy of fruquintinib in neoadjuvant and conversion therapy for locally advanced/advanced colorectal cancer has not yet been reported. This study aims to observe the efficacy and safety of fruquintinib combined with chemotherapy in neoadjuvant or conversion therapy for colorectal cancer patients in the real world.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be enrolled in this study:

  1. Age ≥18 years and ≤75 years;
  2. Either gender;
  3. Patients with histologically confirmed colorectal cancer. For the neoadjuvant treatment cohort: Rectal cancer is limited to high rectal cancer, but patients with mid to low rectal cancer who are unwilling or unsuitable for neoadjuvant chemoradiotherapy can also be included.
  4. Neoadjuvant treatment cohort: Clinically staged as stage II (T3-4N0M0) or stage III (T1-4N1-2M0) and initially resectable; patients with clinical stage M1 but initially resectable can also be included in the neoadjuvant treatment cohort, such as patients with stage IV liver oligometastasis. Conversion treatment cohort: Patients with initially unresectable but potentially resectable locally advanced or advanced distant metastatic colorectal cancer (according to AJCC 8th), and patients with locally advanced low rectal cancer who are unsuitable or unwilling to undergo chemoradiotherapy can also be included.
  5. Have received chemotherapy and fruquintinib for at least 2 cycles. For the neoadjuvant therapy cohort, patients who have not previously received anticancer treatment (radiotherapy, chemotherapy, targeted therapy, or immunotherapy, etc.). The patients are eligible for inclusion in the analysis set if they have received fruquintinib treatment for at least 2 cycles and have undergone at least one tumor assessment after baseline. All patients included in the efficacy analysis are included in the safety analysis set.
  6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 before treatment.
  7. Expected survival time of >6 months before neoadjuvant therapy and >3 months before conversion therapy.
  8. No significant organ dysfunction or drug contraindications before receiving neoadjuvant or conversion therapy.
  9. There is no mandatory requirement for target lesions. Objective response rate (ORR) assessment is based on all evaluable patients, regardless of the presence of target lesions. For patients without target lesions, those assessed as non PR/non PD will be analyzed as stable disease (SD).

Exclusion Criteria:

* Patients meeting any of the following criteria are not eligible to enter the study:

  1. History of other primary malignant tumors, except: (1) complete remission of malignant tumors at least 2 years before enrollment and no need for other treatment during the study period; (2) adequately treated non-melanoma skin cancer or malignant melanoma without evidence of disease recurrence; (3) adequately treated in situ carcinoma.
  2. dMMR/MSI-H.
  3. Female patients who are pregnant or lactating.
  4. Known allergy (Grade 3 or higher allergic reaction) or contraindication to anti-angiogenic drugs or chemotherapy drug components.
  5. Use of non-study drug treatments during the study period that may interfere with the analysis.
  6. Patients who did not undergo any tumor efficacy assessment after receiving neoadjuvant or conversion therapy.
  7. Less than 2 cycles of fruquintinib neoadjuvant or conversion therapy.
  8. Patients with insufficient follow-up information as judged by the investigator (such as not returning to the hospital for treatment or efficacy assessment after initial treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer who have received chemotherapy and fruquintinib as neoadjuvant or conversion treatment.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Corhot1: Pathological Complete Response Rate (pCR) | Time from the first treatment up to 12 weeks
  Pathological Complete Response Rate (pCR), defined as no residual tumor cells in the surgical specimen of the primary tumor and lymph nodes (ypT0N0); corresponds to TRG grade 0.
Corhot2: R0 surgical conversion rate | Time from the first treatment up to 24 weeks
  R0 surgical conversion rate：The proportion of subjects who achieve complete R0 resection of both the primary gastric lesion and any metastases among all subjects receiving the conversion therapy regimen.

SECONDARY OUTCOMES:
Corhot1: R0 resection rate | Time from the first treatment up to 12 weeks
  R0 resection rate: Defined as the proportion of subjects achieving negative margins among those who underwent surgical treatment.
Corhot1: Event-Free Survival (EFS) | Time from the first treatment up to 2 years
  Event-Free Survival (EFS): Time from initiation of neoadjuvant study treatment until first documented progression, recurrence/metastasis, or death from any cause (whichever occurs first, without progression/recurrence at the time of death).
Corhot1: 1-year Event-Free Survival (EFS) rate | Time from the first treatment up to 12 months.
  1-year Event-Free Survival rate: Survival rate of patients who, from initiation of neoadjuvant study treatment, have not experienced progression, recurrence/metastasis, or death from any cause at 12 months.
Corhot1 and Corhot2: Overall Survival (OS) | Time from the first treatment up to 2 years.
  Overall Survival (OS): Time from the first study treatment until death from any cause.
Corhot1 and Corhot2: 1-year Overall Survival (OS) rate | Time from the first treatment up to 12 months.
  1-year OS rate: Survival rate of patients who have not experienced progression or death from any cause at 12 months from the first study treatment.
Corhot1 and Corhot2: Objective Response Rate (ORR) | corhot1 ：Time from the first treatment up to 12 weeks. Corhot2：Time from the first treatment up to 2 years.
  Objective Response Rate (ORR): Proportion of patients with target lesions who achieve a complete response (CR) or partial response (PR) among all treated patients.
Corhot1 and Corhot2: Disease Control Rate (DCR) | corhot1 ：Time from the first treatment up to 12 weeks. Corhot2：Time from the first treatment up to 2 years.
  Disease Control Rate (DCR): Proportion of patients with target lesions who achieve a complete response (CR), partial response (PR), or stable disease (SD) among all treated patients.
Corhot2: Curative Surgery Conversion Rate | Time from the first treatment up to 24 weeks
  Curative Surgery Conversion Rate: The proportion of subjects who undergo potentially curative surgical resection of both the primary gastric lesion and any metastases among all subjects receiving the conversion therapy regimen.
Corhot2: Progression-Free Survival (PFS) | Time from the first treatment up to 2 years.
  Progression-Free Survival (PFS): Defined as the time from initiation of the study treatment regimen until the first radiographic disease progression, postoperative disease recurrence, or death (whichever occurs first). This can be calculated separately for surgical and non-surgical patients, with surgical patients considering postoperative disease recurrence or death (whichever occurs first).
Corhot1and Corhot2: Adverse events | through study completion, an average of 1 year
  Adverse events during neoadjuvant or conversion therapy, impact on surgery (delay, surgical complications) for corhot1, impact on surgical procedure and postoperative outcomes for corhot2.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Xiong, doctor, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No